CLINICAL TRIAL: NCT03999385
Title: Growth and Self-Care: The Use of Mindfulness-Based Interventions to Assist Emerging Adults With Diabetes Transition to Adulthood
Brief Title: Mindful Self-Compassion to Assist Emerging Adults With Diabetes Transition to Adulthood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Michael McIntyre, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H2017:293
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Mindfulness; Mindful Self-compassion; Self-compassion; Diabetes; Self-care
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Pretest-Posttest Waitlist Control Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Training Group (Experimental): 8 weeks of training in Mindful Self-Compassion.
  Interventions: Behavioral: Mindful Self-Compassion (MSC)
- Waitlist Control Group (Other): No intervention for approximately 12 weeks. After this waiting period, participants will complete 8 weeks of training in Mindful Self-Compassion.
  Interventions: Behavioral: Mindful Self-Compassion (MSC)

INTERVENTIONS:
Behavioral: Mindful Self-Compassion (MSC) — The MSC program was developed by Christopher K. Germer, PhD and Kristin Neff, PhD.

SUMMARY:
The transition from pediatric to adult care is particularly difficult for individuals with Type 1 diabetes. It is hypothesized that a mindfulness-based intervention for individuals making this transition will contribute to personal psychological well-being, superior participation in health care, and more tightly controlled blood sugar levels. Young adults with Type I diabetes will complete an eight-week training program in Mindful Self-Compassion. Intervention effectiveness will be assessed with both self-report and physiological measures. Assessments will occur at the start of the training program, end of the program, and three-months post-program.

DETAILED DESCRIPTION:
This research will evaluate the consequences of an eight-week Mindful Self-Compassion (MSC) intervention on the psychological and physical well-being of 18 to 25 year-old individuals with Type 1 diabetes who are at an age of established risk. Participants will be randomly assigned to either an immediate intervention group or wait-list control group. All participants will be tested before and after the intervention on a battery of self-report measures designed to assess various aspects of self-care and psychological functioning. Blood samples will also be taken before and after the intervention to determine HbA1C levels. Participants will also receive a followup assessment three-months post-intervention to assess the durability of the effects. We expect MSC training to induce positive change in participants' diabetes management and personal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 25
* Obtain care for Type 1 diabetes

Exclusion Criteria:

* Psychologically or medically unable to complete the MSC program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in average plasma glucose concentration | Baseline, 8 weeks, and 3 months
  Assessed by HbA1C test results. The desired outcome is a statistically significant decrease in average glucose concentration, indicating greater diabetes management.
Change in diabetes self-management | Baseline, 8 weeks, and 3 months
  Assessed by total scores and subscale scores on the Summary of Diabetes Self-Care Activities (Toobert, Hampson, & Glasgow, 2000), which range from 0 to 7 when item scores are averaged. The items assess general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking. The desired outcome is a statistically significant increase in diabetes self-management.

SECONDARY OUTCOMES:
Change in Self-compassion | Baseline, 8 weeks, and 3 months
  Assessed by total scores and subscale scores on the Self-Compassion Scale (Neff, 2003), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in self-compassion.
Change in Mindfulness | Baseline, 8 weeks, and 3 months
  Assessed by total scores and subscale scores on the Five Facet Mindfulness Questionnaire (Baer et al., 2006), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in mindfulness.
Change in Fears of Compassion | Baseline, 8 weeks, and 3 months
  Assessed by total scores and subscale scores on the Fears of Compassion Scales (Gilbert et al., 2011), which range from 0 to 4 when item scores are averaged. The desired outcome is a statistically significant decrease in fears of compassion.
Change in Positive Affect | Baseline, 8 weeks, and 3 months
  Assessed by total scores on the Positive Affective Well-Being scale (Hess et al., 2005; score range: 1 to 7) and scores on the positive affect subscale of the Positive and Negative Affect Schedule (Watson, Clark, & Tellegen, 1988; score range: 1 to 5). The desired outcome is a statistically significant increase in positive affect.
Change in Negative Affect | Baseline, 8 weeks, and 3 months
  Assessed by scores on the negative affect subscale of the Positive and Negative Affect Schedule (Watson, Clark, & Tellegen, 1988), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant decrease in negative affect.
Change in Perceived Stress | Baseline, 8 weeks, and 3 months
  Assessed by total scores on the Perceived Stress Scale (Cohen et al., 1983), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant decrease in perceived stress.
Change in Life Engagement | Baseline, 8 weeks, and 3 months
  Assessed by total scores on the Life Engagement Test (Scheier et al., 2006), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in life engagement.
Change in Health Locus of Control | Baseline, 8 weeks, and 3 months
  Assessed by subscale scores (internal, chance, powerful others) on the Multidimensional Health Locus of Control Scale (Wallston et al., 1978), which range from 1 to 6 when item scores are averaged. The desired outcome is a statistically significant increase in internal health locus of control.
Change in Eating Disorder Symptomatology | Baseline, 8 weeks, and 3 months
  Assessed by total scores and subscale scores on the Eating Disorders Examination Questionnaire (Fairburn & Beglin, 1994), which range from 0 to 6 when item scores are averaged. The desired outcome is a statistically significant decrease in eating disorder symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McIntyre, Ph.D., Principal Investigator — St. Boniface Hospital Research Centre
Locations (1):
- St. Boniface Hospital Research Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No